CLINICAL TRIAL: NCT04111042
Title: Long-term Outcomes of Colonic Stent as a "Bridge to Surgery" for Malignant Large-bowel Obstruction
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Xavier Serra-Aracil (Unknown); Anna Pallisera-Lloveras (Unknown)
Responsible Party: Principal Investigator, Laura Mora-Lopez, DR, Corporacion Parc Tauli
Other Study IDs: TAULI-STENT
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Stent Occlusion; Long-term Oncologic Results
Keywords: Malignant colonic obstruction; self-expandable metallic stent
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: stenting — stenting procedure in patients diagnosed malignant large bowel occlusion

SUMMARY:
Study of long-term outcomes of colonic stent as a "bridge to surgery" for malignant large-bowel obstruction.

DETAILED DESCRIPTION:
Prospective observational with retrospective analisis study of patients with left-sided malignant colonic obstruction undergoing stenting between April 2006 and April 2018 in Parc Tauli University Hospital. We assessed all patients with intent-to-treat and per protocol analyses in postoperative and long-term follow-up variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years diagnosed with complete malignant colonic obstruction confirmed by CT.
* Elective surgery.
* Location in transverse, left or sigmoid colon.
* Patients who signed the informed consent documentation and agreed to undergo the procedure.

Exclusion Criteria:

* Benign pathology and palliative treatment.
* Unresectable lesion (intraoperative), severe ischemia or cecal perforation, fecal or advanced purulent peritonitis, emergency surgery.
* Previous chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: : patient demographics, physiological status according to the American Society of Anesthesiologist (ASA) score, tumor characteristics and localization, type of surgery, surgical team, stoma formation rate, perioperative morbidity and mortality, tumor stage according to the International Union Against Cancer (UICC)-TNM Classification of Malignant Tumors published by the National Comprehensive Cancer Network (7th edition), administration of adjuvant treatment, local and distant disease recurrence based on CT imaging (and histological tissue if possible), disease-free survival and overall survival.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
long-term outcomes | 2 years
  survival rates

SECONDARY OUTCOMES:
anastomotic leak | 30 days
  surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Mora López, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There's no sharing plan because the study has finished the recruited time